CLINICAL TRIAL: NCT03965117
Title: Effect of Norepinephrine Infusion on Hepatic Blood Flow During Goal-directed Haemodynamic Therapy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019/0395
Record Dates: First submitted 2019-05-20; First posted 2019-05-28 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: General Anesthesia
Keywords: hepatic blood flow; Norepinephrine; hepatic vascular pressure
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- norepinephrine (Experimental): norepinephrine will be started at 0,1 mcg/kg/min and titrated according to its haemodynamic effect.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — norepinephrine will be started at 0,1 mcg/kg/min and titrated according to its haemodynamic effect. After baseline MAP (which is > 60 mmHg), norepinephrine is targeted according baseline MAP. At T2, MAP is between 10 - 20 % above baseline (T1), at T3 MAP is between 20 - 30 % above baseline (T1).

SUMMARY:
Maintaining adequate blood pressure is important for survival of organs. Recent studies have demonstrated that higher blood pressures were necessary for prevention of acute kidney injury and myocardial injury after non-cardiac surgery. Hypotension after induction and maintenance of anesthesia is common. For maintaining adequate blood pressure in a euvolemic patient, vasopressor therapy is required. Norepinephrine (NOR) is commonly used to treat anesthesia-related hypotension.

The hepatic circulation has a large number of alpha and beta adrenergic receptors and is very sensitive for adrenergic stimulation such as norepinephrine infusion. Animal studies (Hiltebrand et al.) suggest that NOR has only minimal effect on hepatic blood flow however the effect of NOR on hepatic blood flow in clinical surgical patients remains unclear.

The aim of the study is to evaluate the effect of NOR on hepatic blood flow during.

goal directed haemodynamic therapy.

DETAILED DESCRIPTION:
All patients receive standardized anesthesia care for pancreas surgery according to the existing departmental protocol for these interventions.

All patients receive individualized goal-directed haemodynamic therapy based on the transpulmonary thermodilution technique.

At designated times, hemodynamic variables will be recorded. These include:

* Heart rate (bpm)
* Central venous pressure (mmHg)
* Mean arterial pressure (mmHg)
* Cardiac index (L/min/m2)
* Pulse pressure variation (PPV)

Blood flow and pressure measurements performed by the surgeon :

* Hepatic flow : hepatic artery (HAF) and portal vein (PVF)
* Pressure measurements in portal vein (PPorta) and caval vein (PCava)

Both flow and pressure will be simultaneously recorded. To minimize the effect of ventilation on pressure, these measurements will be obtained during apnea.

Between each flow measurement there will be a minimum of 5 minutes.

NOR will be started at 0,1 mcg/kg/min and titrated according to its haemodynamic effect. After baseline MAP (which is > 60 mmHg), NOR is targeted according baseline MAP. At T2, MAP is between 10 - 20 % above baseline (T1), at T3 MAP is between 20 - 30 % above baseline (T1).

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years ≤ 80 years (female or male)
* ASA I - II - III
* Able to comprehend, sign and date the written informed consent document to participate in the clinical trial.
* Patient is scheduled for pancreatic surgery.

Exclusion Criteria:

* Allergy to the medication.
* Renal insufficiency (SCr > 2 mg/dL).
* Severe heart failure (EF < 25%).
* Hemodynamic instable patients.
* Atrial fibrillation.
* Sepsis.
* BMI > 40.
* Severe coagulopathy (INR > 2).
* Thrombocytopenia (< 80 x 103 /mcL).
* End stage liver disease.
* Pregnancy and breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
change in hepatic blood flow during goal-directed hemodynamic therapy with norepinphrine | From start anesthesia until end of anesthesia, up to a maximum of 11 hours
  flow measurements with echo probe
change in hepatic blood pressures during goal-directed hemodynamic therapy with norepinphrine | From start anesthesia until end of anesthesia, up to a maximum of 11 hours
  pressure measurements with needle

SECONDARY OUTCOMES:
change in systemic vascular resistance (SVR), during goal-directed hemodynamic therapy with norepinphrine | From start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in systemic vascular resistance (SVR)
change in portal venous resistance (PVR) during goal-directed hemodynamic therapy with norepinphrine | From start anesthesia until end of anesthesia up to a maximum of 11 hours
  change in portal venous resistance (PVR)
change in cardiac index during goal-directed hemodynamic therapy with norepinphrine | From start anesthesia until end of anesthesia, up to a maximum of 11 hours
  change in cardiac index
amount of blood loss | from start of surgery until end of surgery, up to a maximum of 10 hours
  amount of blood loss at end of surgery
amount of fluids given during surgery with goal-directed hemodynamic therapy with norepinphrine | from start of surgery until end of surgery up to a maximum of 10 hours
  total amount of cristalloids and colloids given during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Van Limmen, MD, Principal Investigator — UZ Ghent
Locations (1):
- University Hospital Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Limmen J, Iturriagagoitia X, Verougstraete M, Wyffels P, Berrevoet F, Abreu de Carvalho LF, De Hert S, De Baerdemaeker L. Effect of norepinephrine infusion on hepatic blood flow and its interaction with somatostatin: an observational cohort study. BMC Anesthesiol. 2022 Jul 2;22(1):202. doi: 10.1186/s12871-022-01741-2. PMID 35780092